CLINICAL TRIAL: NCT07140731
Title: An Early Feasibility Study for the Symani Surgical System
Brief Title: The Symani Restore Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jacobs institute (Other)
Responsible Party: Principal Investigator, Adnan Siddiqui, Principal Investigator, Jacobs institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MMI RESTORE CIP-005
Record Dates: First submitted 2025-08-21; First posted 2025-08-26 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Moyamoya Disease
MeSH Terms: conditions — Moyamoya Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single arm study with neurosurgical procedure (Experimental): To assess the safety and effectiveness of the Symani Surgical System
  Interventions: Device: Symani Surgical System

INTERVENTIONS:
Device: Symani Surgical System — To assess the safety and effectiveness of the Symani Surgical System

SUMMARY:
A research study for a neurosurgical procedure in adult patients with Moyamoya disease

DETAILED DESCRIPTION:
The purpose of this research is to assess the safety and effectiveness of the Symani Surgical System in adult patients with Moyamoya disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged >18.
2. Moyamoya disease with minor to moderate symptoms requiring neurosurgical treatment.
3. Patients agree to have the surgery and the anesthesia.
4. Patients who voluntarily decide to participate in this study with the surgery performed with the aid of Symani and agree to sign the Informed Consent Form.

   -

Exclusion Criteria:

1. Patients who have bleeding or coagulation disorders in the past or present.
2. Any criteria that preclude prolonged anesthesia.
3. Hemodynamically unstable neurological exam.
4. Pressure dependent neurologic status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
CT Imaging | 6 Months
  Stable cerebral perfusion confirmed with CT Imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Jacobs Institute, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
Patient privacy